CLINICAL TRIAL: NCT00721214
Title: A Phase II Study of the Use of 5-Azacytidine as Pre-Transplant Cytoreduction Prior to Allogeneic Stem Cell Transplantation for High Risk Myelodysplastic Syndromes
Brief Title: 5-Azacytidine Prior to Allogeneic Stem Cell Transplant in High Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11328
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; 5-azacytidine; allogeneic stem cell transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A: 5-azacytidine (Experimental): 5-azacytidine as pre-transplant cytoreduction prior to allogeneic stem cell transplantation for High Risk Myelodysplatic Syndromes.
  Interventions: Drug: 5-azacytidine

INTERVENTIONS:
Drug: 5-azacytidine — The recommended starting dose for the first treatment cycle, for all patients regardless of baseline hematology laboratory values, is 75 mg/m2 subcutaneously or intravenously, daily for 7 days.
  Other Names: Mylosar; Vidaza; 5-AC; 5-AZC; U-18496

SUMMARY:
The purpose of this study is to examine the feasibility and efficacy of using the demethylating agent 5-Azacytidine prior to allogeneic stem cell transplantation in patients with high risk myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
The study drug, 5-azacytidine, is given daily intravenously for 7 days. After every 2 cycles study participants will have a bone marrow test to evaluate the effect of the 5-azacytidine on the Myelodysplastic Syndrome (MDS). Participants continue to get cycles of 5-Azacytidine until 2 bone marrow tests show the MDS has stopped responding to the treatment. At that time they will undergo a transplant if a donor is available.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the following criteria will be eligible for study entry:

  1. Diagnosis of MDS according to WHO criteria
  2. Intermediate-2 or high risk by IPSS score
  3. Clinically able to receive 5-Azacytidine
  4. Serum bilirubin levels </=1.5 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis
  5. Serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) levels </=2 x ULN
  6. Serum creatinine levels </=1.5 x ULN
  7. Negative serum pregnancy test prior to 5-Azacytidine treatment for women of childbearing potential
  8. Women and men of childbearing potential agree to use contraception while receiving treatment with 5-Azacytidine
  9. Potentially eligible for allogeneic transplantation
  10. No prior allogeneic transplant
  11. Age 18 to 70, inclusive.

Exclusion Criteria:

1. Known or suspected hypersensitivity to 5-azacytidine or mannitol
2. Patients previously treated with 5-azacytidine or deoxyazacytidine
3. Pregnant or breast feeding
4. Patients with advanced malignant hepatic tumors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. McCarty, MD, Study Chair — Virginia Commonwealth University
Locations (1):
- Massey Cancer Center / Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study plans to accrue over one year with a planned 2 year subsequent follow-up. Virginia Commonwealth Unvierstiy (VCU) will be the sole site for this project.
Period: Overall Study
Arm/Group | Arm A: 5-azacytidine
Started | 16
Completed | 12
Not Completed | 4
Not completed — Chose another center for transplant | 1
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: Out of the 16 evaluable patients, 12 were able to proceed to transplant.
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: One Year Overall Survival of Allogeneic Transplant Recipients After Transplantation
Description: Percentage of patients alive one year after their transplantation, as estimated by the Kaplan-Meier survival curve. The estimated one year survival rate from this curve is 50%, while the estimated two year survival rate is 50%.
Time Frame: 1 year
Population: Patients surviving after stem cell infusion will be considered in the transplantation cohort; those dying or relapsing prior to this event are considered to have progressed. Outcomes of 5-Axacytidine responders and non-responders will be compared. Patients alive at the time of last observation will be censored.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 12
percentage of participants | 50 [20 to 80]

2. Secondary Outcome: One-year Overall Survival From Time of Treatment Initiation With 5-Azacytidine for All Study Cohorts
Description: Percentage of participants alive one year after their first treatment was estimated by the Kaplan-Meier survival curve. The events analyzed are evidence of molecular, cytogenetic or histologic relapse or death from any cause. Patients alive at the time of last observation will be censored. The estimated one year overall survival rate from this curve is 47%. The one year overall survival is the same as one year event free survival rate.
Time Frame: 1 year
Population: Intent to treat analysis including patients who consented and were eligible. Patients enrolled in the study having received at least one 28 day cycle of 5-Azacytidine. As well as engraftment of white blood cells and platelets, graft failure, relapse and Graft Versus Host Disease (GVHD) will be considered in the intent-to-treat analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 16
percentage of participants | 47 [20 to 74]

3. Primary Outcome: Two Year Overall Survival of Allogeneic Transplant Recipients After Transplantation
Description: Percentage of patients alive two years after their transplantation, as estimated by the Kaplan-Meier survival curve. The estimated two year survival rate is 50%, the same as one year survival rate.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 12
percentage of participants | 50 [20 to 80]

4. Primary Outcome: One Year Event Free Survival (EFS) for Allogeneic Transplant Recipients After Transplantation
Description: Percentage of participants that received allogeneic transplant and had event free survival, as estimated by the Kaplan-Meier survival curve. The events analyzed are evidence of molecular, cytogenetic or histologic relapse or death from any cause. The estimated one-year event-free survival rate is the same as overall survival, 50%.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 12
percentage of participants | 50 [20 to 80]

5. Primary Outcome: Two Year Event Free Survival (EFS) for Allogeneic Transplant Recipients After Transplantation
Description: Percentage of participants that received allogeneic transplant and had event free survival. The percentage of patients was estimated by the Kaplan-Meier survival curve. The events analyzed are evidence of molecular, cytogenetic or histologic relapse or death from any cause. The estimated two-year event-free survival rate is the same as overall survival, 50%.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 12
percentage of participants | 50 [20 to 80]

6. Secondary Outcome: Two-year Overall Survival From Time of Treatment Initiation With 5-Azacytidine for All Study Cohorts.
Description: Percentage of participants alive two years after their first treatment was estimated by the Kaplan-Meier survival curve. The events analyzed are evidence of molecular, cytogenetic or histologic relapse or death from any cause. Patients alive at the time of last observation will be censored.The estimated two year survival rate is 37% .The estimated two-year overall survival rate is the same as two-year event free survival.
Time Frame: 2 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 16
percentage of participants | 37 [9 to 65]

7. Secondary Outcome: One-year Event-free Survival From Time of Treatment Initiation With 5-Azacytidine for All Study Cohorts
Description: Percentage of participants with one year event free survival after their first treatment was estimated by the Kaplan-Meier survival curve. The events analyzed are evidence of molecular, cytogenetic or histologic relapse or death from any cause. Patients alive at the time of last observation will be censored.The estimated one-year event-free survival rate is the same as for overall survival, 47% (SE = 13.6%).
Time Frame: 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 16
percentage of participants | 47 [20 to 74]

8. Secondary Outcome: Two-year Event-free Survival From Time of Treatment Initiation With 5-Azacytidine for All Study Cohorts
Description: Percentage of participants with two year event free survival after their first treatment was estimated by the Kaplan-Meier survival curve. The events analyzed are evidence of molecular, cytogenetic or histologic relapse or death from any cause. Patients alive at the time of last observation will be censored.The estimated two- year event-free survival rate is the same as for overall survival, 37% (SE = 14.3%).
Time Frame: 2 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 5-azacytidine
Number analyzed (Participants) | 16
percentage of participants | 37 [9 to 65]

ADVERSE EVENTS:
Time Frame: 3 years
Description: Reportable adverse events include relapse, graft failure, any other unexpected grade 3 or 4 that in the opinion of investigator may be related to protocol treatment or death from any cause. All hospitalizations and serious infections (requiring IV antibiotics) will be reported on regular follow-up forms. All other AEs not reportable per protocol.
Arm/Group | Arm A: 5-azacytidine
Serious Adverse Events (participants affected / at risk) | 13/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 5-azacytidine (N=16)
Blood/Bone Marrow - Other (Specify, death-died of progressive MDS) (Blood and lymphatic system disorders) | 4 (4) — Death- died of progressive MDS
Blood/Bone Marrow- Other (Blood and lymphatic system disorders) | 4 (4) — progression/relapse of MDS/AML
Seizure (Nervous system disorders) | 1 (2) — Primary Attribution: Unlikely Detailed Attribution: Other Pt with long history of seizure disorder had single seizure. Was seen in ED and discharged to home
Cholecystitis (Hepatobiliary disorders) | 1 (1) — Primary Attribution: Unrelated Detailed Attribution: Other Drug: 5-Azacytidine Admitted for abdominal pain, found to have acute cholecystitis and had lap cholycystectomy.
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1) — Primary Attribution: Unrelated Detailed Attribution: Other Drug: 5-Azacytidine antibiotics, supportive care Grade 2
Nausea (Gastrointestinal disorders) | 1 (2) — Primary Attribution: Unrelated Detailed Attribution: Other Drug: 5-Azacytidine
Fatigue (Investigations) | 1 (1) — Fatigue (asthenia, lethargy, malaise) Primary Attribution: Unrelated Detailed Attribution: Other Drug: 5-Azacytidine
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dyspnea (shortness of breath) Primary Attribution: Possible Detailed Attribution: Investigational Therapy Drug: 5-Azacytidine
Infection (Blood and lymphatic system disorders) | 1 (1) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Skin (cellulitis) Primary Attribution:Possible Detailed Attribution:Other Drug: 5-Azacytidine
Infection (Blood and lymphatic system disorders) | 2 (2) — Infection with unknown ANC
Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hemorrhage/Bleeding
Opportunistic infection associated with >=Grade 2 Lymphopenia (Blood and lymphatic system disorders) | 1 (1) — patient admitted 3/12/12 for fever and mental status changes, confusion worsened and patient found to have basal ganglia hemorrhage secondary to toxoplasmosis, died in paliative care unit 4/17/12
Died of Sepsis (Infections and infestations) | 3 (3)
Perforation (Gastrointestinal disorders) | 1 (1) — Perforation, GI - Colon
Febrile Neutropenia (Infections and infestations) | 1 (1) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Myositis (Skin and subcutaneous tissue disorders) | 1 (4) — Myositis (inflammation/damage of muscle)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No